CLINICAL TRIAL: NCT02707159
Title: A Novel Therapy for Locally Advanced and Metastatic Pancreatic Cancer Based on Nanoparticle Albumin-bound Paclitaxel and Gemcitabine: Circulating Tumor Cells as a Potential Biomarker for Treatment Monitoring, -Response and Survival
Brief Title: Circulating Tumor Cells as Tools for Therapy Response in Nab-paclitaxel Treated Metastatic Pancreatic Cancer Patients
Acronym: PACT-ACT-v6
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Helse Stavanger HF (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2013/1743; 2013-000633-13 (EudraCT Number)
Record Dates: First submitted 2015-11-22; First posted 2016-03-14 (Estimated); Last update posted 2023-03-08 (Actual); Status verified 2016-03

CONDITIONS: Metastatic Pancreatic Cancer
Keywords: Circulating tumor cells; Nab-paclitaxel; Metastatic pancreatic cancer; Gemcitabine
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplastic Cells, Circulating | interventions — Taxes; Gemcitabine; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nab paclitaxel / gemcitabine (Experimental): Patients will receive 125 mg per m2 nab-paclitaxel and 1000 mg per m2 on days 1, 8 and 15 followed by one week of rest before new treatment cycle.
  Interventions: Drug: Nab paclitaxel / gemcitabine

INTERVENTIONS:
Drug: Nab paclitaxel / gemcitabine — Patients will receive gemcitabine/nab-paclitaxel combination chemotherapy
  Other Names: Nab-paclitaxel and Gemcitabine

SUMMARY:
The majority patients diagnosed with pancreatic cancer have metastatic disease at the time of diagnosis. The prognosis is extremely poor with a 5-year survival rate of less than 5%. Treatment with chemotherapy can improve efficacy, but still the median progression-free survival in patients receiving nab-paclitaxel and gemcitabine is only 5,5 months and median overall survival is less than one year. There is a urgent need for tools for predicting the efficacy of the treatment. The current trial aims at investigating the biomarker potential of circulating tumor cells (CTCs) in metastatic pancreatic cancer patients treated by gemcitabine and nab-paclitaxel.

ELIGIBILITY:
Inclusion Criteria:

* Male or female > 18 years up to 80 years
* Histologically or cytologically proven adenocarcinoma of the pancreas before start of treatment. Also patients for whom there is a strong suspicion of unresectable pancreatic cancer will before the diagnosis is confirmed be asked for consent to take 2 additional biopsies at the time of diagnostic biopsy retrieval, in case the histological analysis confirms that they can be included.
* Locally advanced (primarily unresectable) and/or metastatic disease.
* Presence of at least one measurable lesion according to the RECIST criteria, not restricted to previously irradiated area or limited to bone, pleural effusion or ascites.
* ECOG/WHO performance status ≤2
* Absolute neutrophil count (ANC) >1.5 x 109 /L and platelet count >100 x 109/L
* Total bilirubin < 1.5 times the upper limit of the normal range at the institution (ULN) or AST or ALT < 2 x ULN. If liver metastases are present, patients can be included if total bilirubin < 5× ULN or AST/ALT <10× ULN. Dose reductions of paclitaxel will be performed when bilirubin >2xULN, depending on increase of the bilirubin level according to the recommendations of the Summary of Product Characteristics.
* Serum creatinin < 1,5 ULN / calculated creatine clearance > 60 ml/min.
* Written informed consent

Exclusion Criteria:

* Current infection, bowel obstruction or subobstruction, or other uncontrolled intercurrent illness.
* Prior medical treatment for advanced pancreatic cancer
* Confirmed brain metastasis.
* Concurrent or past history of another malignancy except curatively treated non-melanoma skin cancer or in situ carcinoma of the cervix.
* Treatment with any other investigational drug more than 30 days prior to study entry.
* Allergy to anyone of the included drugs.
* Female patient breast feeding or pregnancy
* Not able/ or not willing to use adequate contraception (defined below). A pregnancy test will be included in the baseline visit for women of childbearing potential.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2014-11; Primary Completion 2017-10 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Change in levels of circulating tumor cells (CTCs) during treatment | Baseline and 9 months

SECONDARY OUTCOMES:
Post-baseline over-all survival | Baseline and 9 months
Post-baseline disease-specific survival | Baseline and 9 months
Post-baseline time to progression | Baseline and 9 months
Clinical response to treatment by RECIST 1.1 | Baseline and 9 months
  Radiologic, clinical and biochemical assessment
Changes in quality of life during treatment | Baseline and 9 months
  Quality of Life is assessed every 4 weeks during treatment and then every 8th weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Bjørnar Gilje, MD, PhD, Principal Investigator — Helse Stavanger HF
Locations (1):
- Stavanger University Hospital, Stavanger, Norway